CLINICAL TRIAL: NCT03634735
Title: Thiamin Against Robust IBD Fatigue
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: TARIF
Record Dates: First submitted 2018-06-11; First posted 2018-08-16 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Fatigue
Keywords: Inflammatory Bowel Disease; Fatigue; Thiamine; Vitamin B1
MeSH Terms: conditions — Fatigue; Inflammatory Bowel Diseases | interventions — Thiamine

STUDY DESIGN:
Intervention Model Description: RCT and crossover
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thiamin (Active Comparator): Oral thiamine: 600 - 1800 mg/day in 4 weeks. Dose is depending on gender and age. Tablet contains 300 mg Thiamine each.
  Interventions: Drug: Thiamine
- Placebo (Placebo Comparator): Placebo: same number of tablets as in the active comparator arm, in 4 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Thiamine — Vitamine B1
  Other Names: Vitamine B1
  Arms: Thiamin
Other: Placebo — Placebo tablets
  Arms: Placebo

SUMMARY:
Patients with Inflammatory Bowel Disease (IBD), disease in remission and chronic fatigue will receive oral Thiamine treatment for 4 weeks in a RCT, cross-over study.

DETAILED DESCRIPTION:
Patients with Inflammatory Bowel Disease (IBD), disease in remission and chronic fatigue will receive high dose oral Thiamine treatment for 4 weeks in a RCT, cross-over study.

After the high dose treatment period, participants will be randomized to 3 months treatment with Thiamine 300mg/day or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Inflammatory Bowel Disease
* Disease in remission
* Chronic fatigue

Exclusion Criteria:

* Co-morbidity that can explain fatigue
* Pregnancy
* Non-compliance to the study procedures
* Possible surgery in the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2020-04-21 (Actual); Study Completion 2020-10-27 (Actual)

PRIMARY OUTCOMES:
Fatigue | After 4 weeks active treatment
  Change in levels of fatigue measured by the Inflammatory Bowel Disease Fatigue Scale (IBD-F). Section I of the scale measures the severity of fatigue on a scale from 0-20, where 20 is maximum fatigue. A change in IBD-F score of 3 points or more is regarded as a clinical relevant change.

SECONDARY OUTCOMES:
Fatigue | Week 8, 12, 24, and 52
  Change in levels of fatigue measured by the Inflammatory Bowel Disease Fatigue Scale (IBD-F). Section I of the scale measures the severity of fatigue on a scale from 0-20, where 20 is maximum fatigue. A change in IBD-F score of 3 points or more is regarded as a clinical relevant change.
Health-Related Quality of Life | Week 4, 8, 12, 24, and 52
  Changes in Health-Related Quality of Life, measured by the generic EQ-5D Tool (mainly the VAS-scale (0-100, where100 is best).
Disease specific Health-Related Quality of Life | Week 4, 8, 12, 24, and 52
  Changes in Health-Related Quality of Life, measured by the disease specific Short Health Scale (SHS). SHS comprises 4 questions regarding disease related quality of life on VAS-scales (0-10, where 10 is worst).

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Central Region, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bager P, Hvas CL, Hansen MM, Ueland P, Dahlerup JF. B-vitamins, related vitamers, and metabolites in patients with quiescent inflammatory bowel disease and chronic fatigue treated with high dose oral thiamine. Mol Med. 2023 Oct 25;29(1):143. doi: 10.1186/s10020-023-00741-3. PMID 37880581
- [Derived] Bager P, Hvas CL, Rud CL, Dahlerup JF. Long-term maintenance treatment with 300 mg thiamine for fatigue in patients with inflammatory bowel disease: results from an open-label extension of the TARIF study. Scand J Gastroenterol. 2022 Jan;57(1):37-43. doi: 10.1080/00365521.2021.1983640. Epub 2021 Sep 30. PMID 34592862
- [Derived] Bager P, Hvas CL, Rud CL, Dahlerup JF. Randomised clinical trial: high-dose oral thiamine versus placebo for chronic fatigue in patients with quiescent inflammatory bowel disease. Aliment Pharmacol Ther. 2021 Jan;53(1):79-86. doi: 10.1111/apt.16166. Epub 2020 Nov 18. PMID 33210299